CLINICAL TRIAL: NCT06102512
Title: A Phase 1, Open-label Two-part Study of the Absorption, Metabolism, Excretion, and the Absolute Bioavailability of [14C]-LOXO-783 in Healthy Adult Subjects
Brief Title: A Study of [14C]-LOXO-783 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-PIK-23005; J4C-OX-JZUE (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [¹⁴C]-LOXO-783 (Part 1) (Experimental): Single dose of [¹⁴C]-LOXO-783 administered orally
  Interventions: Drug: [¹⁴C]-LOXO-783
- LOXO-783 + [¹⁴C]-LOXO-783 (Part 2) (Experimental): Single dose of LOXO-783 administered orally followed by single dose of [¹⁴C]-LOXO-783 administered intravenously (IV)
  Interventions: Drug: LOXO-783; Drug: [¹⁴C]-LOXO-783

INTERVENTIONS:
Drug: [¹⁴C]-LOXO-783 — Administered orally
  Other Names: LY3849524
  Arms: [¹⁴C]-LOXO-783 (Part 1)
Drug: LOXO-783 — Administered orally
  Other Names: LY3849524
  Arms: LOXO-783 + [¹⁴C]-LOXO-783 (Part 2)
Drug: [¹⁴C]-LOXO-783 — Administered IV
  Other Names: LY3849524
  Arms: LOXO-783 + [¹⁴C]-LOXO-783 (Part 2)

SUMMARY:
The main purpose of this study is to evaluate how much of the study drug, the radioactive substance 14C incorporated LOXO-783 ([¹⁴C]-LOXO-783) passes from blood into urine, feces and expired air in healthy adult participants when administered as a single dose. The study will also measure how much of the LOXO-783 and [¹⁴C]-LOXO-783 gets into the bloodstream, how its broken down, and how long it takes the body to get rid of it. The study is conducted in two parts and will last up to approximately 72 and 61 days for part 1 and 2, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants in good health, determined by no clinically significant findings from medical history, physical examination, ECGs, vital signs, and clinical laboratory evaluations as assessed by the investigator
* Have a body mass index within the range 18.5 to 32.0 kilograms per meter squared (kg/m²)
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Fraction of Dose Excreted in Urine (Feur) | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Feur
PK: Cumulative Feur | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Cumulative Feur
PK: Fraction of Dose Excreted in Feces (Fefeces) | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Fefeces
PK: Cumulative Fefeces | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Cumulative Fefeces
PK: Fraction of Dose Excreted in Expired Air (Feair) | Predose on day 1 up to postdose on day 21 (Part 1)
  PK: Feair
PK: Absolute Bioavailability (F) of LOXO-783 | Predose on day 1 up to postdose on day 9 (Part 2)
  PK: F of LOXO-783

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, Study Director — Loxo Oncology, Inc.
Locations (1):
- Fortrea Clinical Research, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No